CLINICAL TRIAL: NCT04538586
Title: Influence of the COVId-19 Pandemic on STRESS, and Screening Procedures
Brief Title: Influence of the COVId-19 Pandemic on STRESS, and Screening Procedures (COVISTRESS Screening)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 COVISTRESS Screening
Record Dates: First submitted 2020-09-03; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: COVID-19 Screening
Keywords: COVID-19; Screening; Stress
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus has caused containment of more than a third of the world's population. Some countries have used a major screening strategy. Screening procedures, such as waiting (or resulting) for the test, can be stressful and can attract the most stressed people. However, there is currently no data on the relationship between stress and screening for SARS-CoV2

DETAILED DESCRIPTION:
This is an observational study by REDCap questionnaire® via a flyer deposited in the waiting room of the COVID screening centres. No incentive to complete the questionnaire will be made. The self-survey will assess stress and its relationship to SARS-CoV2 screening procedures, socio-demographic factors or lifestyle habits. This Screening questionnaire includes 31 questions.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers who are screened

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People screened for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Stress measures | Day 1
  Attitudes and stress related to screening procedure will be measured via questionnaire

SECONDARY OUTCOMES:
Screening | Day 1
  Attitudes towards screening will be measured via questionnaire
Sociodemographic characteristics | Day 1
  Age, gender, qualification, personal work status, ethnicity, life characteristics and stress will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital, Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Delamarre L, Tannous S, Lakbar I, Couarraze S, Pereira B, Leone M, Marhar F, Baker JS, Bagheri R, Berton M, Rabbouch H, Zak M, Sikorski T, Wasik M, Nasir H, Quach B, Jiao J, Aviles R, Covistress Network, Clinchamps M, Dutheil F. The Evolution of Effort-Reward Imbalance in Workers during the COVID-19 Pandemic in France-An Observational Study in More than 8000 Workers. Int J Environ Res Public Health. 2022 Jul 26;19(15):9113. doi: 10.3390/ijerph19159113. PMID 35897478